CLINICAL TRIAL: NCT07164209
Title: Resection of the Mesentery With Functional End-to-end Anastomosis vs Kono Anastomosis in Preventing Relapse After Ileocolic Resection for Primary Crohn Disease: a Prospective, Randomized, Controlled Trial Remeasure CD TRial
Brief Title: The Remeasure Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Ordine Mauriziano di Torino (Other)
Responsible Party: Principal Investigator, Lucia Borsotti, Michela Mineccia, MD, Azienda Ospedaliera Ordine Mauriziano di Torino
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0122316, 14/12/2020
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Ileocolic Crohn Disease; Kono S Anastomosis; Resection of the Mesentery

STUDY DESIGN:
Intervention Model Description: Monocentric, prospective, randomized, controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- resection of the mesentery (Other): Excision of the mesentery:
  the mesentery is fully dissected and excised to the limit of macroscopic "fat wrapping", where mesenteric fat is inflamed and extends beyond its normal anatomical distribution over the surface of the contiguous intestine. The anastomosis between colon and ileum is than performed mechanically end to end
  Interventions: Procedure: Excision of the mesentery: the mesentery is fully dissected and excised to the limit of macroscopic "fat wrapping", where mesenteric fat is inflamed and extends beyond its normal anatomical distribut
- Kono S Anastomosis (Experimental): Kono-S anastomosis:
  the mesentery is not removed but cutted close to the bowel. The bowel is then divided transversely by placing a linear stapler perpendicular to the intestinal lumen and the mesentery. The corners of the two staple lines are reinforced and the two stumps are approximated using 5-7 sutures to create the column.
  If the caliber of the two intestinal segments differs significantly, the sutures should be spaced to evenly distribute the surplus tissue of the larger segment, in order to achieve good approximation and stable support for the anastomosis. To create the anastomosis, an antimesenteric longitudinal enterotomy (or colostomy) is performed on each stump to allow a transverse lumen of 7 cm in diameter for the small bowel or closer to 8 cm for the colon. In this way the supporting column is located immediately behind the posterior wall of the anastomosis providing a rigid and stable support to prevent mechanical deformation and functional constriction of the lum
  Interventions: Procedure: Kono S Anastomosis

INTERVENTIONS:
Procedure: Excision of the mesentery: the mesentery is fully dissected and excised to the limit of macroscopic "fat wrapping", where mesenteric fat is inflamed and extends beyond its normal anatomical distribut — The resection of mesentery could take off the inflammatory tissue who may increase the risk of anastomotic recurrence The Kono anastomosis achieves a column of support (made with the bowel ) located immediately behind the posterior wall of the anastomosis providing a rigid and stable support to prevent mechanical deformation and functional constriction of the lumen of the anastomosis being a barrier between anastomosis and mesentery
  Arms: resection of the mesentery
Procedure: Kono S Anastomosis — ono-S anastomosis: the mesentery is not removed but cutted close to the bowel. The bowel is then divided transversely by placing a linear stapler perpendicular to the intestinal lumen and the mesentery. The corners of the two staple lines are reinforced and the two stumps are approximated using 5-7 sutures to create the column. If the caliber of the two intestinal segments differs significantly, the sutures should be spaced to evenly distribute the surplus tissue of the larger segment, in order to achieve good approximation and stable support for the anastomosis. To create the anastomosis, an antimesenteric longitudinal enterotomy (or colostomy) is performed on each stump to allow a transverse lumen of 7 cm in diameter for the small bowel or closer to 8 cm for the colon. In this way the supporting column is located immediately behind the posterior wall of the anastomosis providing a rigid and stable support to prevent mechanical deformation and functional constriction of the lum
  Arms: Kono S Anastomosis

SUMMARY:
Aim of the present study is to compare a stapled, functional end-to-end, ileo-colic anastomosis with removal of the mesentery vs the manual, functional end-to-end, ileo-colic Kono-S anastomosis with mesentery preservation, in terms of peri-operative safety, and efficacy in preventing endoscopic recurrence after ileocolic resection for Crohn Disease. Patients presenting with ileocolic primary Crohn disease either not suitable for medical treatment or with contraindications for therapy i.e: occlusion, abscess, contraindications to the use of biologics

DETAILED DESCRIPTION:
Patients who meet inclusion criteria will be randomized between two surgical procedures:

The excision of the mesentery (group A) and ileocolic anastomosis and the Kono-S anastomosis (group B) after ileocolic or ileo-cecal resection. The operation could be performed with open or laparoscopic approach.

Excision of the mesentery:

the mesentery is fully dissected and excised to the limit of macroscopic "fat wrapping", where mesenteric fat is inflamed and extends beyond its normal anatomical distribution over the surface of the contiguous intestine. The anastomosis between colon and ileum is than performed mechanically end to end.

Kono-S anastomosis:

the mesentery is not removed but cutted close to the bowel. The bowel is then divided transversely by placing a linear stapler perpendicular to the intestinal lumen and the mesentery. The corners of the two staple lines are reinforced and the two stumps are approximated using 5-7 sutures to create the column.

If the caliber of the two intestinal segments differs significantly, the sutures should be spaced to evenly distribute the surplus tissue of the larger segment, in order to achieve good approximation and stable support for the anastomosis. To create the anastomosis, an antimesenteric longitudinal enterotomy (or colostomy) is performed on each stump to allow a transverse lumen of 7 cm in diameter for the small bowel or closer to 8 cm for the colon. In this way the supporting column is located immediately behind the posterior wall of the anastomosis providing a rigid and stable support to prevent mechanical deformation and functional constriction of the lumen of the anastomosis.

ELIGIBILITY:
Inclusion Criteria:

* • Patients > 18 years

  * Histological diagnosis of Crohn's Disease
  * Patient's ability to read and understand the documentation concerning the study and the Informed consent
  * Ileocolic disease requiring resection

Exclusion Criteria:

* Older than 70

  * Recurrent disease, previous surgery for CD
  * Gastroenterologists or patients not willing to maintain a drug washout for six months
  * Emergency surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
endoscopic recurrence (Rutgeerts score i2 or greater) at 6,12, 18 months.Endoscopic recurrence was defined if Rutgeerts > i2 (>5 aphthous lesions or larger lesions confined to anastomosis), i3 (diffuse ileitis), or i4 (diffuse inflammation with large ulc | From the treatment a close follow up is performed at 6, 12 and 18 months.The majority of endoscopic examinations were centrally performed. In few cases check was performed in separated centers and a "recording video clip" of the endoscopy was assessed fo

CONTACTS AND LOCATIONS:
Locations (1):
- Dott Lucia Borsotti is the head of the experimetal Office in Azienda Sanitaria Ospedaliera Ordine Mauriziano and could answer about enrolling of patients and submission of the protocol to the ethicl Commette of Città della Salute e della Scienza of Torin, Torino, To, Italy

IPD SHARING:
Plan to Share IPD: No
We surely consider to share individual participant data (IPD) during the study and often it is necessary. At the moment of the study design we dis not fix a precise plane of sharing data. During the follow up clinical and endoscopic examinations of patients have been scheduled in order to avoid missing data or drop-out from the study. The first role of all investigators in this study was to follow each patients operated on and enrolled in this specific study

REFERENCES:
- [Background] Coffey CJ, Kiernan MG, Sahebally SM, Jarrar A, Burke JP, Kiely PA, Shen B, Waldron D, Peirce C, Moloney M, Skelly M, Tibbitts P, Hidayat H, Faul PN, Healy V, O'Leary PD, Walsh LG, Dockery P, O'Connell RP, Martin ST, Shanahan F, Fiocchi C, Dunne CP. Inclusion of the Mesentery in Ileocolic Resection for Crohn's Disease is Associated With Reduced Surgical Recurrence. J Crohns Colitis. 2018 Nov 9;12(10):1139-1150. doi: 10.1093/ecco-jcc/jjx187. PMID 29309546
- [Result] Mineccia M, Maconi G, Daperno M, Cigognini M, Cherubini V, Colombo F, Perotti S, Baldi C, Massucco P, Ardizzone S, Ferrero A, Sampietro GM. Has the Removing of the Mesentery during Ileo-Colic Resection an Impact on Post-Operative Complications and Recurrence in Crohn's Disease? Results from the Resection of the Mesentery Study (Remedy). J Clin Med. 2022 Apr 1;11(7):1961. doi: 10.3390/jcm11071961. PMID 35407568
- [Result] Luglio G, Rispo A, Imperatore N, Giglio MC, Amendola A, Tropeano FP, Peltrini R, Castiglione F, De Palma GD, Bucci L. Surgical Prevention of Anastomotic Recurrence by Excluding Mesentery in Crohn's Disease: The SuPREMe-CD Study - A Randomized Clinical Trial. Ann Surg. 2020 Aug;272(2):210-217. doi: 10.1097/SLA.0000000000003821. PMID 32675483

DOCUMENTS (2):
  • Study Protocol (2025-09-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT07164209/Prot_000.pdf
  • Informed Consent Form (2025-09-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT07164209/ICF_001.pdf